CLINICAL TRIAL: NCT03082105
Title: Evaluation of Air Pocket Factors That Contribute to the Development of Hypoxia and Hypercapnia
Brief Title: Snow Physical Properties and Human Ventilatory Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: V/16/13
Record Dates: First submitted 2017-03-08; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Hypoxic Respiratory Failure; Hypercapnic Respiratory Failure; Avalanche Burial; Snow Physical Properties
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiration; Snow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Winter snow (Experimental): First test series breathing in dry snow in winter
  Interventions: Other: Breathing in snow
- Intermediate snow (Experimental): Second test series breathing in dry/wet snow in intermediate season
  Interventions: Other: Breathing in snow
- Spring snow (Experimental): Third test series breathing in very wet snow in spring
  Interventions: Other: Breathing in snow

INTERVENTIONS:
Other: Breathing in snow — Breathing in snow with different physical properties

SUMMARY:
Sufficient oxygenation is critical for completely buried avalanche victims to avoid life-threatening consequences during hypoxic exposure. Snow contains a remarkable capacity to maintain air availability; it was suspected that the snow physical properties affect the development of hypoxia and hypercapnia. The aim of this study was to evaluate the influence of different snow physical properties on the development of hypoxia and hypercapnia in subjects breathing into an artificial air pocket in snow. Twelve male healthy subjects breathed through an airtight face-mask and 40cm tube into an artificial air pocket of 4L. Every subject performed three tests on different days with varying snow characteristics. Symptoms, gas and cardiovascular parameters were monitored up to 30min. Tests were interrupted at SpO2 <75% (primary endpoint); or due to subjective symptoms like dyspnea, dizziness, and headache (i.e. related to hypercapnia). Snow density was assessed via standard methods and micro-computed tomography (CT) analysis, and permeability and penetration with the snow micro-penetrometer (SMP).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with an age above 18yr-old, physically active.
* Volunteers have been informed and have signed consent.

Exclusion Criteria:

* Lack of consent.
* Chronic previous illness of the respiratory tract or of the cardiovascular system.
* Acute disease at or immediately prior to the test (eg, flu-like infection, fever of unknown origin).
* Eurac employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-03-09 (Actual); Study Completion 2014-03-09 (Actual)

PRIMARY OUTCOMES:
SpO2 (%) | Changes from baseline (measurement at 0min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption of snow-breathing phase [max 30min]) -> 2.5min and 5min after snow-breathing phase
  Continuous monitoring

SECONDARY OUTCOMES:
EtCO2 (mmHg) | Changes from baseline (measurement at 0min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption of snow-breathing phase [max 30min]) -> 2.5min and 5min after snow-breathing phase
  Continuous monitoring
Cause of interruption | Timepoint immediately before interruption of snow-breathing phase (max 30min)
  SpO2 <75% or subjectives symptoms due to hypercapnia (like dyspnea, dizziness, and headache)
VE (L/min) | Changes from baseline (measurement at 0min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption of snow-breathing phase [max 30min]) -> 2.5min and 5min after snow-breathing phase
  Continuous monitoring
rSO2 (%) | Changes from baseline (measurement at 0min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption of snow-breathing phase [max 30min]) -> 2.5min and 5min after snow-breathing phase
  Continuous monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Strapazzon, MD PhD, Study Director — Eurac Research; Hermann Brugger, MD, Study Director — Eurac Research
Locations (1):
- Institute of Mountain Emergency Medicine, Eurac Research, Bolzano, Bz, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brugger H, Sumann G, Meister R, Adler-Kastner L, Mair P, Gunga HC, Schobersberger W, Falk M. Hypoxia and hypercapnia during respiration into an artificial air pocket in snow: implications for avalanche survival. Resuscitation. 2003 Jul;58(1):81-8. doi: 10.1016/s0300-9572(03)00113-8. PMID 12867313
- [Background] Haegeli P, Falk M, Brugger H, Etter HJ, Boyd J. Comparison of avalanche survival patterns in Canada and Switzerland. CMAJ. 2011 Apr 19;183(7):789-95. doi: 10.1503/cmaj.101435. Epub 2011 Mar 21. PMID 21422139